CLINICAL TRIAL: NCT05072457
Title: Benefit of Assistive Listening Device for Lateralization and Spatial Hearing
Brief Title: Benefit of Assistive Listening Device for Lateralization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Hearts for Hearing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SRF-387
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-05

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental (Experimental): All participants in the study fit with Phonak Audeo P hearing aids and compatible Phonak Roger receivers.
  Interventions: Device: Roger On microphone; Device: Roger Select microphone

INTERVENTIONS:
Device: Roger On microphone — Roger On microphone transmitter which is used with Roger receivers and Audeo P hearing aids
Device: Roger Select microphone — Roger Select microphone transmitter which is used with Roger receivers and Audeo P hearing aids

SUMMARY:
Speech intelligibility in noise will be evaluated in adults with moderate to moderate-severe sensorineural hearing loss using a Phonak Roger microphone and hearing aid with compatible Phonak Roger receiver. Target speech will be presented from multiple directions while competing diffuse background noise is presented simultaneously. Participants will repeat back words and percent correct is calculated.

ELIGIBILITY:
Inclusion Criteria:

* Experienced hearing aid users, age 18 or older
* Bilateral, symmetric moderate to moderate-severe sensorineural hearing loss
* Good understanding of the English language
* Health outer ear as confirmed by otoscopy
* Informed consent as documented by signature

Exclusion Criteria:

* Contraindications to the medical device noted upon otoscopy
* Known hypersensitivity or allergies to materials of the investigations device or comparator
* Inability to produce reliable test results
* Known psychological problems
* Self reported symptoms of vertigo or dizziness

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-07-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hearts for Hearing, Oklahoma City, Oklahoma, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adults with moderate-severe bilateral sensorineural hearing loss
Arm/Group | Experimental
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 74 [48 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Lateralization Hearing Ability
Description: Participants indicate which direction (left, center, or right) target speech sentences are coming from while competing noise is also presented via four corner speakers. A higher number of correct responses indicates better lateralization ability. This will be done with two Roger microphone systems (Roger On and Roger Select)
Time Frame: Day 1 of 1 day study
Measure: Mean (Full Range); unit: percent correct responses
Arm/Group | Experimental
Number analyzed (Participants) | 10
percent correct responses
  % Correct using Roger On microphone | 71 [53.33 to 100]
  % Correct using Roger Select microphone | 54 [26.67 to 73.33]
Statistical Analysis 1: Comparison: Experimental; MANOVA analysis with independent variable being the intervention condition (type of microphone used) and dependent variable being the performance on lateralization task. Null hypothesis: There will be no statistically significant difference in lateralization test scores between the Roger On and the Roger Select in the experimental group; Test type: Other; p < .05, ANOVA

2. Primary Outcome: Spatial Hearing Ability
Description: Participants repeat sentences presented from the left speaker, while ignoring overlapping competing sentences presented from the right speaker. A higher percentage of correctly repeated words indicates a better spatial hearing score. This task will be performed using two Roger microphone systems (Roger On and Roger Select)
Time Frame: Day 1 of 1 day study
Measure: Mean (Full Range); unit: percentage of words correctly repeated
Arm/Group | Experimental
Number analyzed (Participants) | 10
percentage of words correctly repeated
  % Correct using Roger On microphone | 48 [7.78 to 72.5]
  % Correct using Roger Select microphone | 42 [5.1 to 73.75]
Statistical Analysis 1: Comparison: Experimental; Independent variable: intervention condition (type of microphone used), Dependent variable: performance on spatial hearing task. Null hypothesis: There will be no statistically significant difference in spatial hearing test scores between the Roger On and the Roger Select in the experimental group; Test type: Other; p > .05, ANOVA

ADVERSE EVENTS:
Time Frame: 1 day
Description: All participants underwent testing with both the Roger On Microphone and the Roger Select Microphone during one day testing session. Therefore, all participants are combined for the Adverse Event Reporting.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT05072457/Prot_SAP_000.pdf